CLINICAL TRIAL: NCT06603545
Title: The Effect of Digital Education for Osteoporosis Patients on Fracture Risk and Related Health Outcomes in Older Swedish Men and Women.
Brief Title: The Effect of Digital Education for Osteoporosis Patients on Fracture Risk and Related Health Outcomes.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Uppsala University Hospital (Other); Region Stockholm (Other Government); Västernorrland County Council, Sweden (Other Government); Region Västerbotten (Other Government); Region Skane (Other); Norrbottens Lans Landsting (Other)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Senior Consultant in Geriatric Medicine, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEOP001
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoporosis; Accidental Falls; Fractures, Bone; Patient Reported Outcome Measures; Drug Adherence; Injury Traumatic
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Medication Adherence; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital education for osteoporosis patients (DEOP) (Experimental): The participants in the DEOP group will be given access to the DEOP for four months after randomization, and can redo the education multiple times within those four months. Reminders will be sent out using phone text messages monthly for the first 3 months to participants who have not yet started the DEOP.
  The experimental group will also be given information, according to standard care, regarding fall prevention, physical activity, diet, and osteoporosis medication according to standard care, by their GP or the physician at the osteoporosis clinics, depending on where they are treated for their osteoporosis.
  Interventions: Other: Digital education for osteoporosis patients
- No Digital education for osteoporosis patients (DEOP) (No Intervention): The control group will be given information regarding fall prevention, physical activity, diet, and osteoporosis medication according to standard care, by their GP or the physician at the osteoporosis clinics, depending on where they are treated for their osteoporosis.

INTERVENTIONS:
Other: Digital education for osteoporosis patients — DEOP is found on the Swedish health care system's dedicated website or app 1177, it takes approximately 60 minutes to complete and is composed of three modules: 1)Introduction: an animated video that shows the patient flow from having a fracture, being evaluated at the osteoporosis clinic, receiving information about osteoporosis, and being treated for osteoporosis. 2)Osteoporosis: basic information about osteoporosis; why it occurs, risk factors that the patient can affect (such as physical inactivity and smoking), and risk factors that cannot be affected (such as age and heredity). It provides information about typical osteoporotic fractures, and how a patient is evaluated according to clinical guidelines for osteoporosis care. 3)Treatment: information about the different kinds of pharmacological osteoporosis treatment, physical activity, balance control, lifting technique, risk of falling, and dietary advice, especially regarding calcium and vitamin D intake.
  Other Names: DEOP
  Arms: Digital education for osteoporosis patients (DEOP)

SUMMARY:
A digital education for osteoporosis patients (DEOP) has been developed and tested on patients in Region Vastra Gotaland, Sweden. Currently, the evidence regarding the efficacy of patient education on fracture risk, medication adherence, injurious falls, levels of physical activity, and diet is insufficient. Most patients with osteoporosis in Sweden are diagnosed and treated in primary care, where the knowledge about osteoporosis is often very limited. Thus, in general, osteoporosis patients are not sufficiently informed before receiving a treatment recommendation. This randomized controlled trial aims to investigate if DEOP vs. standard care can reduce the incidence of fracture in older women and men, and if the intervention leads to better adherence to osteoporosis medication, higher quality of life, increased physical activity, and enhanced diet.

The primary objective is to investigate if DEOP compared to standard care (without DEOP), can reduce the incidence of clinical fractures in men and women, over the age of 65 years, without previous osteoporosis medication the last year, who have been recommended osteoporosis treatment after a DXA scan and assessment of clinical risk factors at an osteoporosis clinic.

The secondary objectives are to investigate if DEOP compared to standard care (without DEOP), can reduce the incidence of injurious falls, have positive effects on adherence to osteoporosis medication, positively affect diet (calcium and vitamin D intake), physical activity, and improve quality of life in men and women, over the age of 65 years, without previous osteoporosis medication the last year, who have been recommended osteoporosis treatment after a DXA scan and assessment of clinical risk factors at an osteoporosis clinic.

Study design: randomized multicentre clinical trial. Patients over the age of 65 visiting an osteoporosis unit for a bone density scan (DXA) will be asked to participate in the study. The participants will be randomized to one of two arms where one arm will be invited to DEOP and the other arm will receive standard care, without DEOP.

DETAILED DESCRIPTION:
The hypothesis is that improved patient education using an easily accessible online educational material will result in better adherence to osteoporosis medication and positive lifestyle changes, which will lead to a lower risk of fractures and injurious falls. The primary aim of this study is to investigate if a Digital Education for Osteoporosis Patients (DEOP) affects the risk of sustaining a clinical fracture in patients over the age of 65 who have been recommended osteoporosis treatment after a bone density (DXA) scan. The secondary aims are to investigate if DEOP affects the risk of injurious falls, adherence to osteoporosis medications, improves dietary intake and quality of life, and increases physical activity compared to standard care.

The planned study is a multicentre randomized controlled trial, with 9 participating study centers (osteoporosis clinics). Patients who have not previously received osteoporosis medication the last year and are over the age of 65 visiting an osteoporosis clinic for a clinical evaluation, including a bone density scan (DXA) and assessment of clinical risk factors and fracture risk, will be asked to participate in the study. Before the appointment for the DXA measurement, possible study participants will receive written information about the study by mail. At the visit, oral information about the study will be provided by the bone densitometry technologist. Written information will be distributed to possible participants that have not previously received the information. The patients must have the opportunity to ask questions before they make their decision to participate or not. Acceptance to participate must be communicated both verbally and through signing an informed consent form. All patients will undergo a DXA-scan and answer a questionnaire regarding clinical risk factors included in the fracture risk assessment tool FRAX, according to local clinical guidelines.

At a later stage, if the patient, by the doctor at the osteoporosis clinic, is recommended pharmacological treatment for osteoporosis (due to a high fracture risk), the patient becomes eligible for the study. If the patient does not have an indication to receive osteoporosis medication, as judged by the physician at the osteoporosis unit, the patient will be excluded from the study as screening failure and receive a notification of this through e-mail or regular mail.

Patients eligible for the study will be randomized, stratified according to sex and study center, into one of two arms where patients in one arm will be invited to the DEOP and patients in the other arm will receive standard care, without the DEOP. Patients in both groups will be treated and followed according to clinical guidelines for osteoporosis care in their health care region, by either a general practitioner (GP) or a doctor at an osteoporosis clinic. Only osteoporosis clinics without an ongoing DEOP will be eligible as study clinics in these health care regions. After randomization, the local study coordinator will contact all included patients through e-mail or regular mail and ask them to complete self-reported questionnaires regarding physical activity, diet, and quality of life (Physical Activity Scale for the Elderly (PASE), Food Frequency Questionnaire (FFQ), and quality of life (Short Form survey, SF-12), respectively). Data regarding clinical risk factors (and calculated 10-year probability of major osteoporotic fracture and hip fracture) in the fracture risk assessment tool FRAX, height, and weight, and bone mineral density (BMD; of the lumbar spine, total hip, and femoral neck, in grams/cm2 and as T-scores) will be collected from the osteoporosis clinic by the local study coordinator or other study personnel. After years 1 and 3, an e-mail or regular mail (if the study participant does not use e-mail) will be sent to the participants and they will be asked to answer the same questionnaires again. Data regarding clinical fractures will be collected from the Patient Register (Socialstyrelsen, the National Board of Health and Welfare), the Swedish Fracture Register, and from regional X-ray archives after the end of the study (maximum 4 years of follow-up). Data on the incidence of injurious falls (including injuries without fracture) will be collected through the Patient Register at the end of the study. Data on osteoporosis medication use will be collected from the Drug Dispensation Register and regional databases regarding medications provided at health care facilities at the end of the study. Data on deaths will be collected using the National Cause of Death Register. Data on diagnoses and medication will be collected five years back from the inclusion date to determine comorbidity.

The participants in the DEOP group will be given access to the DEOP for four months after randomization. Reminders will be sent out using phone text messages monthly for the first 3 months to participants who have not yet started the DEOP. The control group will be given information regarding fall prevention, physical activity, diet, and osteoporosis medication according to standard care, by their GP or the physician at the osteoporosis clinics, depending on where they are treated for their osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting an osteoporosis unit, 65 years and older.
* Ability to understand and follow study instructions.
* Signed informed consent.
* Have been recommended pharmacological osteoporosis treatment after a clinical evaluation including a DXA-scan and assessment of fracture risk at an osteoporosis clinic.
* Have access to www.1177.se.

Exclusion Criteria:

* Patients with previous osteoporosis medication the last year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2640 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Time to first event of clinical fracture. | Maximum follow-up four years.
  Time to first event of clinical fracture.

SECONDARY OUTCOMES:
Time to event death. | Maximum follow-up four years.
  Time to event death.
Time to first event of an injurious fall | Maximum follow-up four years.
  Time to first event of an injurious fall
Adherence (percent remaining on treatment) to osteoporosis drug therapy at years 1 and 3. | At years 1 and 3.
  Adherence (percent remaining on treatment) to osteoporosis drug therapy at years 1 and 3.
Change in physical activity level from randomization to years 1 and 3. | From randomization to years 1 and 3.
  Change in physical activity level, measured in the Physical Activity Scale of the Elderly (PASE; 0-793) from randomization to years 1 and 3.
Change in dietary intake (total daily intake of calcium and vitamin D) from randomization to years 1 and 3. | From randomization to years 1 and 3.
  Change in dietary intake (total daily intake of calcium (mg/day) and vitamin D (IU/day)) from randomization to years 1 and 3.
Change in quality of life from randomization to years 1 and 3. | From randomization to years 1 and 3.
  Change in quality of life (measured using the SF-12 scale) from randomization to years 1 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorentzon, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: No